CLINICAL TRIAL: NCT06025942
Title: Enhancing Emotion Regulation With an In-situ Socially Assistive Robot Among LGBTQ+ Youth With Self-harm Ideation: a Randomised Control Trial
Brief Title: Purrble With LGBTQ+ Youth Who Have Self-harmful Thoughts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: University of Oxford (Other); University of Nottingham (Other); University of Glasgow (Other); Stanford University (Other); University of Melbourne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RESCM-22/23-34570
Record Dates: First submitted 2023-08-29; First posted 2023-09-06 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-03

CONDITIONS: Emotion Regulation; Self Harm
Keywords: LGBTQ; Self-harm; Emotion regulation; Young people; RCT
MeSH Terms: conditions — Emotional Regulation; Self-Injurious Behavior

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): The Purrble intervention takes the form of an interactive plush toy, designed to be handed over to the young person and support in-the-moment soothing.
  Interventions: Behavioral: Purrble intervention
- Control (No Intervention): Wait-list control (access to services as usual)

INTERVENTIONS:
Behavioral: Purrble intervention — When the Purrble is picked up, it emits a frantic heartbeat that slows down if the person uses calm stroking movements. If the Purrble is soothed for long enough, it transitions into a purring vibration indicating a calm, content state.
  Logic model underlying the intervention:
  Level 1: in-the-moment soothing support to young people in emotional moments when they would attempt to utilise emotion regulation (ER) strategies to calm down.
  Level 2: mechanisms that facilitate long-term engagement with the intervention, building on positive subjective experience of Level 1.
  Level 3: shift in young peoples' ER practices and implicit beliefs about emotion, after repeated experience of Levels 1-2.
  * see JMIR Res Protoc 2021;10(11):e28914 (doi: 10.2196/28914)
  Arms: Intervention

SUMMARY:
The primary aim of the proposed Randomised Control study is to investigate the effects of a socially assisted robot (i.e. Purrble) on emotional regulation difficulties (measured by DERS8) with young LGBTQ+ people who have self-harmful (with or without suicidal intention) (in comparison to a wait-listed control).

Secondary aims include investigating the effects of the Purrble on young people's self-harmful thoughts, symptoms of anxiety and depression, alongside quantitative and qualitative (interviews) measures of engagement with the intervention.

DETAILED DESCRIPTION:
Self-harm is a key concern among young people, this is highlighted by the rising rates self-harm and suicide attempts in recent years. Internationally, young LGBTQ+ people are recognised to report higher prevalence of self-harmful thoughts, behaviours, anxiety and depression than their cisgender, heterosexual peers. Emotion regulation (ER) is known to be a transdiagnostic risk factor, which is widely associated with higher risk of self-harm. Typically, LGBTQ+ populations also report greater difficulties with ER which partially explains association with self-harm.

While LGBTQ+ youth are frequent users of digital technologies and digital interventions are often considered feasible and acceptable, there is limited evidence of the effectiveness of such within these populations. Currently, there is no evidence-based digital interventions targeting LGBTQ+ youth who struggle with self-harm.

To address this gap, the investigators have conducted a small pilot study (n=21) to evaluated one such possible tool - Purrble - as a means to offer in-the-moment emotional support for those with high levels of self-harm risk (high symptoms of anxiety, depression, or self-harmful experiences in the last 6 months). The goals of the study centre around testing the feasibility, acceptability, and usage of Purrble across a 2-week deployment period. These results have been promising, indicating Purrble as a feasible and acceptable intervention, alongside indicators of clinical value during Purrble deployment: i) reduction of anxiety and depression symptoms during deployment and ii) reduced prevalence of self-harm thoughts.

From previous interviews, participants highlighted the positive outcomes which were associated with Purrble use (stopping them reaching the point of thinking about self-harm, being a barrier to self-harm behaviours, and encouraging emotional regulation coping strategies; e.g. grounding, self-soothing). However, these pilot studies did not include a controlled waitlist group, and thus more rigorous investigation of these promising effects is needed - leading to the current study.

ELIGIBILITY:
Inclusion Criteria:

Currently experiencing self-harmful thoughts (within the last month) Identify as sexual orientation or gender identity minority (LGBTQ+) Aged 16-25 years Currently living in the UK at the time of the study Able to read and write in English

Exclusion Criteria:

Young people who live outside the UK, are not within the 16-25 year age bracket, and are not experiencing self-harmful thoughts will not be included in the study.

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 155 (Actual)
Dates: Start 2024-01-11 (Actual); Primary Completion 2024-10-23 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Emotion regulation (DERS8) | all timepoints [Time Frame: Three times during pre-deployment (week 1-3) and ten times during the 10-week long deployment period (week 4-13) = total of 13 times]
  Across the trial, we hypothesise that access to the Purrble intervention (compared to the waitlist control) will lead to a decrease in self-reported difficulties with emotion regulation as measured by the primary outcome (DERS8). We will compare the DERS8 assessment pre-deployment (calculated as the average of DERS scores across baseline weeks 1-3) and final deployment assessments (averaged across weeks 11-13).
  Measured by: Difficulties with Emotional Regulation Scale-8 (DERS8), an 8-item instrument used to measure or assess the difficulties with regulating emotion [22].
  The DERS8 score is calculated using a 5-point Likert scale, ranging from 1 (almost never, 0-10%) to 5 (almost always 91-100%). These scores are added together to form a total score (8-40). Higher scores indicate greater levels of difficulty associated with response to situations eliciting negative emotions.

SECONDARY OUTCOMES:
Self-harmful thoughts (SHQ) | all timepoints [Time Frame: Three times during pre-deployment (week 1-3) and ten times during the 10-week long deployment period (week 4-12) = total of 13 times]
  A secondary aim to evaluate the impact of the Purrble intervention on young LGBTQ+ people's self-harmful ideation (with and without suicidal intention), compared to waiting list controls.
  Measured by: The Self-Harm Questionnaire (SHQ; [23]). While the whole instrument is used at baseline (T0), offering a greater level of detail as to why someone has self-harmed, and only the three screener items will be used across deployment. These question the presence of self-harmful thoughts (without suicidal intentions), suicidal thoughts, and whether the young person has harmed themselves on purpose. The screener assigns scores of 1 (no), 2 (yes, once), 3 (yes, two, three or four times), and 4 (yes, five or more times) - offering a general idea of frequency of self-harmful thoughts.
Anxiety (GAD7) | all timepoints [Time Frame: Three times during pre-deployment (week 1-3) and ten times during the 10-week long deployment period (week 4-13) = total of 13 times]
  A secondary aim is to investigate the effects of Purrble on reports of anxiety symptoms within young LGBTQ+ people who have current experiences of self-harmful ideation (in comparison to a wait-listed group).
  Measured by: Generalised Anxiety Disorder Assessment (GAD-7; [24]), a seven-item instrument that is used to measure or assess the severity of generalised anxiety disorder. Each item asks the individual to rate the severity of their symptoms over the past two weeks.
  The GAD-7 score is calculated by assigning scores of 0, 1, 2, and 3, to the response categories of "not at all," "several days," "more than half the days," and "nearly every day," respectively, and then adding together the scores for the seven questions (score range: 0-21). Scores of 5, 10, and 15 represent cut-points for mild, moderate, and severe anxiety, respectively.
Depression (PHQ-9) | all timepoints [Time Frame: Three times during pre-deployment (week 1-3) and ten times during the 10-week long deployment period (week 4-13) = total of 13 times]
  A secondary aim is to investigate the effects of Purrble on reports of depressive symptoms within young people who have current experiences of self-harmful ideation (in comparison to a wait-listed group).
  Measured by: Patient Health Questionnaire-9 (PHQ-9; [25]) , a depression module which scores each of the nine DSM-IV criteria as "0" (not at all) to "3" (nearly every day). It is not a screening tool for depression but it is used to monitor the severity of depression and response to treatment. The maximum score is 27 (9 questions x maximum 3 points per question). Depression severity is graded based on the PHQ-9 score: None 0-4 Mild 5-9 Moderately 10-14 Moderately severe 15-19 Severe 20-27.

OTHER OUTCOMES:
Emotion regulation (PMERQ) | 3 timepoints [Timeframe: Once during pre-deployment (week 3 [T0]) and twice during the 10 -week long deployment period (week 8 [T5], week 13 [T10]) = total of 3 times]
  An additional aim is to examine the levels of endorsement for attentional deployment among LGBTQ+ youth; we hypothesise that those with access to Purrble will score higher than those in the waitlist control.
  Measured by: The Process Model of Emotion Regulation Questionnaire (PMERQ; [26]), a 45-item measure which considers 10 ER strategies across the five stages of the Process Model of ER, and particularly how these strategies are used to decrease negative emotions. A Likert-scale is used, scoring 1 (strongly disagree) to 6 (strongly agree).
  We only include 2 subscales which focus on attention deployment (focusing elsewhere - 4-items (4-24) and cognitive distraction 5-items (5-30)). Each subscale is scored by taking the average of item-level responses, with higher scores indicating greater endorsement.
Hopefulness (SHS) | [Timeframe: Once during pre-deployment (week 3 [T0]) and twice during the 10 -week long deployment period (week 8 [T5], week 13 [T10]) = total of 3 times]
  An additional aim is to examine the levels of hope among LGBTQ+ youth; we hypothesise that those with access to Purrble will score higher than those in the waitlist control.
  Measured by: The State Hope Scale (SHS; [27]) is a 6-item self-report measure of ongoing goal-directed thinking (agency and pathways). Responses are rated on an 8-point Likert scale ranging from 1 (Definitely True) to 8 (Definitely False) with higher scores indicative of greater state hopefulness (total score: 6-48).
Loneliness (UCLA) | 3 timepoints [Timeframe: Once during pre-deployment (week 3 [T0]) and twice during the 10 -week long deployment period (week 8 [T5], week 13 [T10]) = total of 3 times]
  An additional aim is to examine the levels of loneliness among LGBTQ+ youth; we hypothesise that those with access to Purrble will score lower than those in the waitlist control.
  The UCLA Loneliness scale for children [28]) is a 3-item measure used to assess loneliness using 3 responses; 1 (hardly ever or never), 2 (some of the time), and 3 (often). Scores range from 3-12, with higher scores indicating greater levels of loneliness.
Engagement with the Purrble intervention (TWEETS) | all timepoints following deployment for intervention group [Time frame: Ten times during the 10-week long deployment period (week 4-13)]
  An additional aim includes investigating the engagements with the Purrble over the 10-week deployment period among intervention participants.
  Measured by: Measured by: An adapted version of Twente Engagement with eHealth Technologies Scale (TWEETS; [29]). Consisting of 9-items measured on a 5-point Likert scale ranging from strongly disagree (0) to strongly agree (4), total score ranging from 0-36. Engagement is split into subsections considering behaviour, cognitive and affective engagement. Higher scores indicate greater engagement with the intervention.
Engagement with the Purrble intervention | all timepoints following deployment for intervention group [Time frame: Ten times during the 10-week long deployment period (week 4-13)]
  An additional aim includes investigating the engagements with the Purrble over the 10-week deployment period among intervention participants.
  Measured by: A bespoke survey informed by the previous Purrble research [30]. The questions inquire about Purrble use and perceived usefulness. Items are rated on a 0 to 4 scale unless otherwise specified.
  How often did participants engage with Purrble this week? If not at all, why do participants think that was? On average, did engaging with Purrble make any difference to how participants felt at the time?

CONTACTS AND LOCATIONS:
Locations (1):
- King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Data will be available upon reasonable request once the trial is complete. To date there is no data that has been collected or analysed for this study. The data will be held at King's College London, following the data management agreement of Digital Youth.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Access to the data will be available once the trial is complete. Trial end date is currently September 2025
Access Criteria: Reasonable requests for access to the data will be reviewed by core study team

REFERENCES:
- [Background] Gillies D, Christou MA, Dixon AC, Featherston OJ, Rapti I, Garcia-Anguita A, Villasis-Keever M, Reebye P, Christou E, Al Kabir N, Christou PA. Prevalence and Characteristics of Self-Harm in Adolescents: Meta-Analyses of Community-Based Studies 1990-2015. J Am Acad Child Adolesc Psychiatry. 2018 Oct;57(10):733-741. doi: 10.1016/j.jaac.2018.06.018. Epub 2018 Aug 21. PMID 30274648
- [Background] Griffin E, McMahon E, McNicholas F, Corcoran P, Perry IJ, Arensman E. Increasing rates of self-harm among children, adolescents and young adults: a 10-year national registry study 2007-2016. Soc Psychiatry Psychiatr Epidemiol. 2018 Jul;53(7):663-671. doi: 10.1007/s00127-018-1522-1. Epub 2018 May 2. PMID 29721594
- [Background] Coker TR, Austin SB, Schuster MA. The health and health care of lesbian, gay, and bisexual adolescents. Annu Rev Public Health. 2010;31:457-77. doi: 10.1146/annurev.publhealth.012809.103636. PMID 20070195
- [Background] Haas AP, Eliason M, Mays VM, Mathy RM, Cochran SD, D'Augelli AR, Silverman MM, Fisher PW, Hughes T, Rosario M, Russell ST, Malley E, Reed J, Litts DA, Haller E, Sell RL, Remafedi G, Bradford J, Beautrais AL, Brown GK, Diamond GM, Friedman MS, Garofalo R, Turner MS, Hollibaugh A, Clayton PJ. Suicide and suicide risk in lesbian, gay, bisexual, and transgender populations: review and recommendations. J Homosex. 2011;58(1):10-51. doi: 10.1080/00918369.2011.534038. PMID 21213174
- [Background] Marshal MP, Dietz LJ, Friedman MS, Stall R, Smith HA, McGinley J, Thoma BC, Murray PJ, D'Augelli AR, Brent DA. Suicidality and depression disparities between sexual minority and heterosexual youth: a meta-analytic review. J Adolesc Health. 2011 Aug;49(2):115-23. doi: 10.1016/j.jadohealth.2011.02.005. Epub 2011 May 26. PMID 21783042
- [Background] Saewyc EM. RESEARCH ON ADOLESCENT SEXUAL ORIENTATION: DEVELOPMENT, HEALTH DISPARITIES, STIGMA AND RESILIENCE. J Res Adolesc. 2011 Feb 15;21(1):256-272. doi: 10.1111/j.1532-7795.2010.00727.x. PMID 27099454
- [Background] McDermott E, Hughes E, Rawlings V. Norms and normalisation: understanding lesbian, gay, bisexual, transgender and queer youth, suicidality and help-seeking. Cult Health Sex. 2018 Feb;20(2):156-172. doi: 10.1080/13691058.2017.1335435. Epub 2017 Jun 23. PMID 28641479
- [Background] Irish M, Solmi F, Mars B, King M, Lewis G, Pearson RM, Pitman A, Rowe S, Srinivasan R, Lewis G. Depression and self-harm from adolescence to young adulthood in sexual minorities compared with heterosexuals in the UK: a population-based cohort study. Lancet Child Adolesc Health. 2019 Feb;3(2):91-98. doi: 10.1016/S2352-4642(18)30343-2. Epub 2018 Dec 12. PMID 30552054
- [Background] Chan MK, Bhatti H, Meader N, Stockton S, Evans J, O'Connor RC, Kapur N, Kendall T. Predicting suicide following self-harm: systematic review of risk factors and risk scales. Br J Psychiatry. 2016 Oct;209(4):277-283. doi: 10.1192/bjp.bp.115.170050. Epub 2016 Jun 23. PMID 27340111
- [Background] Sloan E, Hall K, Moulding R, Bryce S, Mildred H, Staiger PK. Emotion regulation as a transdiagnostic treatment construct across anxiety, depression, substance, eating and borderline personality disorders: A systematic review. Clin Psychol Rev. 2017 Nov;57:141-163. doi: 10.1016/j.cpr.2017.09.002. Epub 2017 Sep 11. PMID 28941927
- [Background] Wolff JC, Thompson E, Thomas SA, Nesi J, Bettis AH, Ransford B, Scopelliti K, Frazier EA, Liu RT. Emotion dysregulation and non-suicidal self-injury: A systematic review and meta-analysis. Eur Psychiatry. 2019 Jun;59:25-36. doi: 10.1016/j.eurpsy.2019.03.004. Epub 2019 Apr 12. PMID 30986729
- [Background] Fox KR, Franklin JC, Ribeiro JD, Kleiman EM, Bentley KH, Nock MK. Meta-analysis of risk factors for nonsuicidal self-injury. Clin Psychol Rev. 2015 Dec;42:156-67. doi: 10.1016/j.cpr.2015.09.002. Epub 2015 Sep 12. PMID 26416295
- [Background] Kapatais A, Williams AJ, Townsend E. The Mediating Role of Emotion Regulation on Self-harm among Gender Identity and Sexual Orientation Minority (LGBTQ+) Individuals. Arch Suicide Res. 2023 Apr-Jun;27(2):165-178. doi: 10.1080/13811118.2022.2064254. Epub 2022 Apr 21. PMID 35446245
- [Background] Fraser G, Wilson MS, Garisch JA, Robinson K, Brocklesby M, Kingi T, O'Connell A, Russell L. Non-Suicidal Self-Injury, Sexuality Concerns, and Emotion Regulation among Sexually Diverse Adolescents: A Multiple Mediation Analysis. Arch Suicide Res. 2018 Jul-Sep;22(3):432-452. doi: 10.1080/13811118.2017.1358224. Epub 2017 Sep 7. PMID 28759324
- [Background] Steinke J, Root-Bowman M, Estabrook S, Levine DS, Kantor LM. Meeting the Needs of Sexual and Gender Minority Youth: Formative Research on Potential Digital Health Interventions. J Adolesc Health. 2017 May;60(5):541-548. doi: 10.1016/j.jadohealth.2016.11.023. Epub 2017 Jan 17. PMID 28108088
- [Background] Bowen D, Jabson J, Kamen C. mHealth: an avenue for promoting health among sexual and gender minority populations? Mhealth. 2016 Sep 19;2:36. doi: 10.21037/mhealth.2016.09.01. eCollection 2016. No abstract available. PMID 28293609
- [Background] Strauss P, Morgan H, Wright Toussaint D, Lin A, Winter S, Perry Y. Trans and gender diverse young people's attitudes towards game-based digital mental health interventions: A qualitative investigation. Internet Interv. 2019 Sep 5;18:100280. doi: 10.1016/j.invent.2019.100280. eCollection 2019 Dec. PMID 31890628
- [Background] Gilbey D, Morgan H, Lin A, Perry Y. Effectiveness, Acceptability, and Feasibility of Digital Health Interventions for LGBTIQ+ Young People: Systematic Review. J Med Internet Res. 2020 Dec 3;22(12):e20158. doi: 10.2196/20158. PMID 33270039
- [Background] Penner F, Steinberg L, Sharp C. The Development and Validation of the Difficulties in Emotion Regulation Scale-8: Providing Respondents with a Uniform Context That Elicits Thinking About Situations Requiring Emotion Regulation. J Pers Assess. 2023 Sep-Oct;105(5):657-666. doi: 10.1080/00223891.2022.2133722. Epub 2022 Oct 28. PMID 36306434
- [Background] Ougrin D, Boege I. Brief report: the Self Harm Questionnaire: a new tool designed to improve identification of self harm in adolescents. J Adolesc. 2013 Feb;36(1):221-5. doi: 10.1016/j.adolescence.2012.09.006. Epub 2012 Oct 6. PMID 23046733
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Olderbak S, Uusberg A, MacCann C, Pollak KM, Gross JJ. The Process Model of Emotion Regulation Questionnaire: Assessing Individual Differences in Strategy Stage and Orientation. Assessment. 2023 Oct;30(7):2090-2114. doi: 10.1177/10731911221134601. Epub 2022 Dec 9. PMID 36495015
- [Background] Snyder CR, Sympson SC, Ybasco FC, Borders TF, Babyak MA, Higgins RL. Development and validation of the State Hope Scale. J Pers Soc Psychol. 1996 Feb;70(2):321-35. doi: 10.1037//0022-3514.70.2.321. PMID 8636885
- [Background] Kelders SM, Kip H, Greeff J. Psychometric Evaluation of the TWente Engagement with Ehealth Technologies Scale (TWEETS): Evaluation Study. J Med Internet Res. 2020 Oct 9;22(10):e17757. doi: 10.2196/17757. PMID 33021487
- [Derived] Williams AJ, Cleare S, Borschmann R, Tench CR, Gross J, Hollis C, Chapman-Nisar A, Naeche N, Townsend E, Slovak P; Digital Youth. Enhancing emotion regulation with an in situ socially assistive robot among LGBTQ+ youth with self-harm ideation: protocol for a randomised controlled trial. BMJ Open. 2024 Jan 9;14(1):e079801. doi: 10.1136/bmjopen-2023-079801. PMID 38195171